CLINICAL TRIAL: NCT05338164
Title: Protective Value of Cervical Cerclage Against Preterm Birth in Twin Pregnancy With Short Cervix. A Randomized Controlled Trial.
Brief Title: Prophylactic Cerclage for Twin Pregnancy With Shortened Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZU-IRB #8090/17-10-2021
Record Dates: First submitted 2021-12-11; First posted 2022-04-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Preterm Birth; Twin Pregnancy With Antenatal Problem; Cervical Shortening
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerclage group (Experimental): cervical cerclage between 14 and 20 weeks will be done by one of the three authors.
  Interventions: Procedure: cervical cerclage
- No Cerclage group (No Intervention): Routine follow up without cerclage

INTERVENTIONS:
Procedure: cervical cerclage — McDonald cervical cerclage will be applied using Mersaline braided tape with double needle. Single stitch (4 bites) will be applied as close as possible to the level of internal os. The Knot will be put either anterior or posterior according to the surgeon desire.
  Arms: Cerclage group

SUMMARY:
This randomized controlled trial is aimed to evaluate pregnancy and neonatal outcomes in twin pregnancies, in which a cervical cerclage is placed due to the shortening of the cervix with or without visible fetal membranes.

DETAILED DESCRIPTION:
Introduction Multiple pregnancies are high-risk pregnancies and usually associated with an increased risk of neonatal morbidity and mortality, mainly due to preterm births. Preterm births occur in 50% of twin pregnancies and the mean gestational age for delivery is 35.3 weeks. Ten percent of all twin births take place before 32 weeks of gestation.1 Preterm births are responsible for more than 70% of all neonatal and infant mortality.2 Prematurity can have serious consequences for the child, such as hearing difficulties, vision impairment, learning disabilities, reduced IQ, and cerebral palsy. A cervical length of ≤25 mm in twin pregnancies is a good predictor of a spontaneous preterm birth when measured around 24 weeks of gestation.3,4 Numerous interventions have been attempted in order to prevent preterm births in twin gestations, but until now, no intervention has been effective. Use of cerclage in twin pregnancies is controversial. Some experts claim that placing a cervical cerclage could increase the risk of preterm births.5 However, there is growing evidence of beneficial effect of applying cervical cerclage. Based on a few, small, controlled trials, cervical cerclage may extend the pregnancy, if it is applied to a cervix of less than 15 mm.6,7 Such practice is still in need for further validation by well-structured and powered randomized controlled trials.

Rationale:

Pregnant in twins with history suggesting cervical weakness and evidence of shortened cervix in the current pregnancy might get benefit from mechanical support by cervical cerclage in trial to reduce the risk of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years.
* Dichorionic twins.
* Transvaginal sonographic cervical length is <25 mm with or without internal os dilatation ≥10 mm at 14-20 weeks gestational age.
* Asymptomatic.

Exclusion Criteria:

* Triplets and quadruplets.
* Monochorionic twins.
* Threatened/ inevitable miscarriage
* Bulging membranes through the external os.
* Extremes of age.
* Major fetal anomalies.
* Known cases with uterine anomalies e.g. bicornuate uterus, uterus didelphis… etc.
* Fetal demise.
* Fetal reduction in the current pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant ladies
Enrollment: 100 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The incidence of preterm birth at ≤33+6, and ≤31+6 weeks with cervical length ≤25 mm | Immediate reporting of cases at time of delivery through study completion, an average of 1 year
  Rate of preterm births stratified by gestational age inside the included women

SECONDARY OUTCOMES:
Subgroup analysis for the risk of preterm birth at ≤33+6, and ≤31+6 weeks with cervical length ≤15 mm | Immediate reporting of cases at time of delivery through study completion, an average of 1 year
  subgroup analysis for rate of preterm births for very short cervix
The incidence of miscarriage. | Immediate reporting of cases at time of miscarriage through study completion, an average of 1 year
  rate of missed, inevitable and complete miscarriages
Incidence of cervico-vaginal infection | after confirmation of infection through study completion, an average of 1 year
  Rate of infections diagnosed during pregnancy by patient complaint, clinical examination and confirmed by culture and sensitivity).
Neonatal outcomes in both groups | early neonatal through study completion, an average of 1 year
  Rate of untoward early neonatal outcomes respiratory distress, IVH, necrotizing enterocolitis, sepsis, NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Lashiin, M.D., Principal Investigator — Zagazig University; Amro El Nemr, M.D., Principal Investigator — Zagazig University
Locations (1):
- Faculty of medicine, Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No